CLINICAL TRIAL: NCT03225417
Title: Phase Ib/II Trial to Evaluate Safety and Efficacy of Oral Ixazomib in the Prophylaxis of Chronic Graft-versus-host Disease.
Brief Title: Ixazomib in the Prophylaxis of Chronic Graft-versus-host Disease.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X16082
Record Dates: First submitted 2017-04-04; First posted 2017-07-21 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Hematopoietic Stem Cell Transplantation; Multiple Myeloma
Keywords: Ixazomib
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Tacrolimus; Sirolimus; Cyclophosphamide; In Vitro Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Phase I: Ixazomib + Tacrolimus + Sirolimus. Ixazomib doses in this study is 3 to 4 mg of ixazomib on day +1, +8 and +15. Tacrolimus at a dose of 0.02 mg/kg/day and then 0.06 mg/kg/day. Sirolimus at a dose of 6 mg on day -5 and then 4 mg per day.
  Phase II: Ixazomib+ any prophylaxis for GVHD, except antithymocyte globulin, cyclophosphamide or any T depletion protocol in vitro or in vivo.
  Starting Dose of Ixazomib according to phase I.
  Interventions: Drug: Ixazomib; Drug: Tacrolimus; Drug: Sirolimus; Drug: Any prophylaxis for GVHD
- Control group (Other): Any prophylaxis for GVHD, except antithymocyte globulin, cyclophosphamide or any T depletion protocol in vitro or in vivo.
  Interventions: Drug: Tacrolimus; Drug: Sirolimus; Drug: Any prophylaxis for GVHD

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules. Phase I: Starting dose of Ixazomib: 3.0 or 4.0 mg by day +1, +8 and +15. Phase II: Starting Dose of Ixazomib: Maximum tolerated dose from Phase I.
  Other Names: X16082
  Arms: Experimental group
Drug: Tacrolimus — Tacrolimus at dose of 0.02 mg/kg/day and then 0.06 mg/kg/day.
  Other Names: Prograf
Drug: Sirolimus — Sirolimus oral solution. Standing 6 mg orally on day -5 and continued 4mg per day. This drugs should be slowly tapered starting 3 months posttransplant in order to stop them at 9 to 12 months posttransplant according to physician criteria.
  Other Names: Rapamune
Drug: Any prophylaxis for GVHD — Except antithymocyte globulin, cyclophosphamide or any T depletion protocol in vitro or in vivo.
  Other Names: Any prophylaxis for GVHD, except antithymocyte globulin, cyclophosphamide or any in vitro or in vivo.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HTC) is the only curative option for many patients with hematologic malignancies but >50% of this patients will develop extensive chronic graft-versus-host disease (cGVHD), which remains the most important complication after HTC.

Classically, the most effective strategies to prevent GVHD have not improved survival; therefore, the new strategies are being sought.

This study is designed in two phases: the main objective for phase I study is the more suitable dose for ixazomib search. Phase II study is designed to evaluate the efficacy of ixazomib at the doses stablished in phase I.

DETAILED DESCRIPTION:
The study design is based on a phase I / II trial in eight Spanish hospitals.

In the phase I, a number of 3 to 12 patients will be included to evaluate the optimal dose of ixazomib in combination with sirolimus and tacrolimus.

In the phase II, a total number of 130 patients will be randomized to receive ixazomib or the best medical recommendation added in order to evaluate the efficacy of ixazomib. This patients who will receive any prophylaxis for GVHD, except those patients who received antithymocyte globulin , cyclophosphamide or any T depletion protocol in vitro or in vivo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older.
2. Patients on the day +100 +/- 20 days who have received an allogeneic transplant with myeloablative or reduced intensity conditioning peripheral blood allogeneic stem cell transplantation.
3. Patients who have received a hematopoietic bone marrow transplant hematopoietic progenitors of peripheral blood from histo / compatible donor as definition accepted by protocol.
4. Patients receiving any prophylaxis for GVHD, except for antithymocyte globulin, cyclophosphamide or any in vitro or in vivo depletion protocol.
5. Voluntary written consent must be given before performance of any study related procedure.
6. Female patients who accomplish with requisitions for not possibility of pregnancy (menopausal, effective methods of contraception), as detailed by protocol.
7. Eastern Cooperative Oncology Group performance status and/or other performance status 0, 1, or 2.
8. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count 1,000/mm3 and platelet count 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
   * Total bilirubin 1.5 the upper limit of the normal range .
   * Alanine aminotransferase and aspartate aminotransferase 3 upper limit of the normal range.
   * Calculated creatinine clearance 30 mL/min.
9. Ability to swallow and tolerate oral medication.
10. Absence of gastrointestinal symptoms that precludes oral intake and absorption.
11. Off antibiotics and amphotericin B formulations, voriconazole or other anti-fungal therapy for the treatment of active proven, probable or possible infections.
12. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Major surgery within 14 days before enrollment.
3. Central nervous system involvement with malignant cells.
4. Uncontrolled infection within 14 days before study enrollment.
5. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
6. Systemic treatment, within 14 days before the first dose of ixazomib, with strong Cytochrome P450, family 3, subfamily A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
7. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus positive.
8. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
9. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
10. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
11. Patient has Grade 1 with pain or ≥ grade 2 with or without pain peripheral neuropathy.
12. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
13. Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not.
14. Active Graft versus host disease at the time of inclusion: patients are allowed to be included if acute Graft-versus-host Disease is in complete remission and are receiving systemic steroids at < 0.25 mg / kg.
15. Active hematologic malignancy at the time of inclusion.
16. Active microangiopathy at the time of inclusion (according to International Working Group criteria).
17. Gastrointestinal disease or procedure than can interfere with oral absorption , intolerance to the ixazomib or difficulty to swallow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximun tolerated dose | 3 months after transplantation (a total of 3 cycles of 28 days length of study treatment)
  Maximun tolerated dose of the ixazomib in combination with sirolimus and tacrolimus in patients following allogeneic stem cell transplantation for the phase I study will be determinated
Efficacy of ixazomib for phase II study | 9 months after transplantation (a total of 9 cycles of 28 days length of study treatment)
  Presence of moderate plus severe Chronic Graft-versus-host Disease according to NIH scale in patients receiving the maximum tolerated dose.

SECONDARY OUTCOMES:
Event immune recovery for the phase I study | The post-transplant days +180, +270, +365, +545, +730
  Quantification of time of event immune recovery in patients exposed and not exposed to ixazomib.
Event free survival for phase II study. | Just after the time of transplantation and 1 and 2 years after transplantation
  Quantification of time of event free survival for patients receiving the maximum tolerated dose.
Event immune recovery for phase II study. | The post-transplant days +180, +270, +365, +545, +730
  Quantification of time of event immune recovery in patients exposed and not exposed to ixazomib.
Exposure to immunosuppressive treatment for phase II study. | 1 and 2 years after transplantation.
  Evaluation of needs of additional permitted immunosuppressive treatment administered as concomitant medication
Overall disease free survival for phase II study | 2 years after transplantation.
  Quantification of time of overall survival after study treatment
Serious adverse event for phase II study | 1 and 2 years after transplantation
  Describe the serious adverse event notified during the study
Risk of moderate or severe GVHD for phase II study | 2 years after transplantation
  To evaluate the risk of moderate or severe GVHD according to the NIH scale
Differences among patients receiving a reduced-intensity and myeloablative conditioning regimen for phase II study. | 1 and 2 years after transplantation
  To evaluate differences in terms of chronic GVHD and treatment tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Antonio Perez-Simon, MD-PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (8):
- Spain (8):
  - ICO- Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall D´Hebrón, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico Universitario Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data for primary and secondary variables is planned to be shared with all participants within 6 months of data completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after data completion
Access Criteria: Investigators participating in the study until the final publication is done

REFERENCES:
- [Derived] Caballero-Velazquez T, Delgado Serrano J, Lopez-Corral L, Ferra-Coll C, Garcia-Calderon CB, Valcarcel D, Garcia-Cadenas I, Perez Lopez E, Jimenez Lorenzo MJ, Martin-Dominguez FM, Jimenez-Leon MLR, Orti G, Escamilla Gomez V, Blazquez-Goni C, Cabero Martinez A, Andrade Ruiz H, Menendez-Pedregal E, Sanchez-Guijo F, Perez Simon JA. Ixazomib decreases the risk of chronic graft-versus-host disease: identification of cGVHD biomarkers. Blood Adv. 2025 Nov 11;9(21):5528-5538. doi: 10.1182/bloodadvances.2025016284. PMID 40737543